CLINICAL TRIAL: NCT04099134
Title: PaCaReg: A Multicenter Registry Trial for the Assessement of Clinical, Epidemiological and Biological Profiles in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: PACAREG: a Multicenter Registry Trial in Pancreatic Ductal Adencarcinoma
Acronym: PaCaReg
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Head of department for internal medicine I, University of Ulm
Other Study IDs: PaCaReg
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Pancreas Adenocarcinoma; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * Tumor tissue from biopsies or surgery
  * Blood samples at defined timepoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PaCaReg is a multicenter registry trial aiming in the assessement of clinical, epidemiological and biological profiles in patients with pancreatic ductal adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive histologically or cytologically proven pancreatic ductal adenocarcinoma (PDAC) or highly suspicious diagnosis (only pre-curative-intended resection)
* Age =>18 years
* written informed consent

Exclusion Criteria:

* papillary cancer
* neuroendocrine pancreatic tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult newly diagnosed patients with a PDAC could be included in the registry trial.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
General assessment of applied therapy modalities in pancreatic cancer | First diagnose to death or end of surveillance (5 years after curative resection)
Quality of life in pancreatic cancer patients | First diagnose to death or end of surveillance (5 years after curative resection)
  EORTC QLQ c30 and PAN 26

SECONDARY OUTCOMES:
General epidemiologic assessment | First diagnose to death or end of surveillance (5 years after curative resection)
  Epidemiologic questionaire
Assessment of tumor surveillance in pancreatic cancer patients | First diagnose to death or end of surveillance (5 years after curative resection)
Evaluation of predictive and prognostic markers | First diagnose to death or end of surveillance (5 years after curative resection)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, MD, Principal Investigator — Ulm University Hospital
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany